CLINICAL TRIAL: NCT01694524
Title: Nervous System Infections Among Patients With Febrile Seizure : Retrospective Cohort Review of Consecutive Patients Admitted in 7 Pediatric Emergency Departments in Ile-de-France Between 2007 and 2011
Brief Title: Nervous System Infections Among Patients With Febrile Seizure
Status: Completed | Type: Observational
Sponsor: Hôpital Armand Trousseau (Other)
Collaborators: Hopital Universitaire Robert-Debre (Other); Hôpital Jean Verdier (Other); Centre Hospitalier Intercommunal Creteil (Other); Versailles Hospital (Other); Centre hospitalier Lagny Marne la vallée (Unknown); Centre hospitalier intercommunal de Poissy (Unknown)
Responsible Party: Principal Investigator, CARBAJAL, Professor, Hôpital Armand Trousseau
Other Study IDs: febrile seizure and infection
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Seizure; Febrile Seizure; Meningitis; Encephalitis
MeSH Terms: conditions — Seizures; Seizures, Febrile; Meningitis; Encephalitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Few studies dealing with the risk of infectious of nervous system and the utility of lumbar puncture and of emergent neuroimaging among patients with simple febrile seizure between 3 and 11 months age and with complex seizure has been reported. None of these studies was multicentric. Recommendations about management of these children are heterogeneous.

The investigators aim to study by an observational retrospective multicentric study the rate of infectious of central nervous system among patients with a complex febrile seizure and among patients between 3 and 11 months age with simple febrile seizure.

ELIGIBILITY:
Inclusion Criteria:

* febrile (>38°)
* Seizure

Exclusion Criteria:

* previous non febrile seizure
* known trauma
* immunodeficiancy status
* Underlying illness

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This was a retrospective cohort review of consecutive patients admitted in 7 pediatric emergency departments in Ile-de-France between 2007 and 2011. All clinically well-apparent children 3 to 11 months of age with a first simple febrile seizure were included in the study. All children between 3 months and 5 years with a complex febrile seizure were included
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Bacterial meningitis | 7 days after emergency visit
  Results of lumbar puncture or meningitis history in charts
Herpes simplex virus meningitis/encephalitis | 7 days after emergency visit
  Results of lumbar puncture or meningitis history in charts

SECONDARY OUTCOMES:
emergent intracranial processus | 7 days after emergency visit

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Carbajal, MD, PhD, Principal Investigator — Hôpital Armand Trousseau, Paris
Locations (7):
- France (7):
  - Hopital Jean Verdier, Bondy
  - Centre hospitalier intercommunal de creteil, Créteil
  - Centre hospitalier Lagny-Marne la Vallée, Lagny-sur-Marne
  - Centre hospitalier de Versailles, Le Chesnay
  - Hôpital Armand Trousseau, Paris
  - Hopital Robert Debré, Paris
  - Centre hospitalier intercommunal de Poissy, Poissy